CLINICAL TRIAL: NCT02590406
Title: EPO2-A: Evaluation of Different Pre-Oxygenation Condition in Morbid Obesity: Effect of Position and Positive Pressure Ventilation During General Anesthesia Induction
Brief Title: EPO2-A: Evaluation of Pre-Oxygenation in Morbid Obesity: Effect of Position and Positive Pressure Ventilation
Acronym: EPO2-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IUCPQ 21211
Record Dates: First submitted 2015-10-06; First posted 2015-10-29 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Obesity, Morbid
Keywords: Morbid Obesity; Bariatric Surgery; Pre-Oxygenation; Anesthesia Induction; Positive pressure ventilation; Non hypoxic apnea time; Positive-Pressure Respiration; Anesthesia, General
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beach chair (BC) and ZEEP (Active Comparator): Table Position: Beach chair, Inclination of the upper part of the table at 25 degrees, breaking at the patient's hips ZEEP: 3 minutes pre-oxygenation with tidal volumes, FiO2 100%, mouth piece used as a ventilatory interface
  Interventions: Procedure: Beach chair (BC) and ZEEP
- Reverse Trendelenburg and NIPPV (Experimental): Table Position: Reverse Trendelenburg, Inclination of the whole table at 25 degrees from an horizontal plane, head up.
  NIPPV: 3 minutes of pre-oxygenation with 8 cm H2O positive pressure and 10 cm H2O PEEP. Trigger set at 1,5 L/min, mouth piece is used as a ventilatory interface
  Interventions: Procedure: Reverse Trendelenburg and NIPPV

INTERVENTIONS:
Procedure: Beach chair (BC) and ZEEP — Table Position: Beach chair, Inclination of the upper part of the table at 25 degrees, breaking at the patient's hips ZEEP: 3 minutes pre-oxygenation with tidal volumes, FiO2 100%, mouth piece used as a ventilatory interface
  Arms: Beach chair (BC) and ZEEP
Procedure: Reverse Trendelenburg and NIPPV — Table Position: Reverse Trendelenburg, Inclination of the whole table at 25 degrees from an horizontal plane, head up.
  NIPPV: 3 minutes of pre-oxygenation with 8 cm H2O positive pressure and 10 cm H2O PEEP. Trigger set at 1,5 L/min, mouth piece is used as a ventilatory interface
  Arms: Reverse Trendelenburg and NIPPV

SUMMARY:
The risk of complication associated with airway in obese patient is important. The result of pre-oxygenation gives the clinician a prolonged non-hypoxic apnea time. The relation between FRC and non-hypoxic apnea time has been correlated. However, the best condition to accomplish the pre-oxygenation in morbidly obese patient has yet to be described in the medical literature. A study previously done in our hospital (EPO2-PV) compared the effect of different positions and ventilation modes on the FRC in the laboratory. A significant difference has been established on the FRC between the inverse Trendelenburg position with positive pressure ventilation and the head up ("beach-chair") position without positive pressure. The current study, EPO2-A is designed to compared the two positions and ventilation modes during the induction of general anesthesia on morbidly obese and correlate the difference in FRC to difference in apnea time.

DETAILED DESCRIPTION:
Obesity prevalence in the population is increasing. Thus a growing number of obese patient need surgical interventions. These patients have a four time higher risk of suffering of serious complication in relation with their airway management compare with non-obese patients. This is explained by an increased incidence of difficulty with the ventilation and intubation of the obese. The time available for the clinician to manage the airway is define by the non hypoxic apnea time. This laps of time is dependent of the oxygen stocks of the patient, which are dependent of the functional residual capacity (FRC) and his oxygen consumption. For a non-obese patient, a normal pre-oxygenation of three minutes at 100% of oxygen allows a non hypoxic apnea time (oxygen saturation > 90%) of 8,9 minutes. However, for the morbidly obese, this time is cut to less than three minutes.

The major goal of the pre-oxygenation is to increase the alveolar partial pressure of oxygen available in the end-expiratory pulmonary volume. This can be done by replacing the nitrogen in the alveolus by oxygen and by increasing the pulmonary stocks, the FRC. It has been demonstrated that the FRC after the induction of anesthesia is cut by half for the obese. This reduction is explained by a diminished thoracic compliance and an increase of the dependent lung regions' atelectasis because of a more cephalic position of the diaphragm.

Various pre-oxygenation methods have been described to prolong the non hypoxic apnea time in the obese population. Some proposed pre-oxygenation strategies with the patient in the head up position (beach chair). It is a position derived from the ramped position described as the best to visualized the obese patients' glottis. Others proposed pre-oxygenation strategies with positive pressure ventilation, but only the supine position has been studied concomitantly.

Individually, these techniques of pre-oxygenation are superior to the combination of supine position and no positive pressure. Indeed, studies demonstrated that the beach chair position (derived from the ramped position) or the positive pressure pre-oxygenation in supine position diminished the time needed to obtain a satisfactory pre-oxygenation (End-expiratory oxygen fraction >0,9) and a longer non hypoxic apnea time. Sill, these strategies have never been combined in the same protocol.

The beach chair position without positive pressure ventilation has become the standard of care because it is the position that allows the best glottis view. Though, it has been shown by Boyce and coll. that the reverse Trendelenburg position, and not the beach chair, increased the non hypoxic apnea time, the recuperation time and the minimal saturation obtained compared to the supine position. We think that there is an advantage to use the reverse Trendelenburg position to optimize the non hypoxic apnea time. Indeed, our hypothesis is that there will be less pressure on the diaphragm in comparison with the beach char position.

A studied realized by our group (EPO2-PV) evaluated the effect of three positions (Reverse Trendelenburg, beach chair and supine) and two ventilation strategies (spontaneous ventilation with or without positive pressure) on morbidly obese FRC in laboratory. The results showed a statistically significant difference on the FRC after a pre-oxygenation with positive pressure compared with the pre-oxygenation without positive pressure, and this regardless of the position. Moreover, for both ventilation strategies, results demonstrated a statistically significant superiority between the FRC obtained after pre-oxygenation in reverse Trendelenburg compared with the beach chair and the supine position. No improvement has been shown with the beach chair position.

Thereby, the current study will try to correlate the FRC results obtained in laboratory in actual non hypoxic apnea time in the operating room. This research design tries to compare, in patient receiving general anesthesia for bariatric surgeries, the effect of the pre-oxygenation with positive pressure and the reverse Trendelenburg position, on the non hypoxic apnea time in comparison with the actual standard of care, beach chair position without positive pressure ventilation.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40
* Abdominal obesity : waist circumference: > 115 for the women waist circumference > 130 for the men

Exclusion Criteria:

* Facial hair
* Cranio-facial abnormality
* Asthma (continuous treatment)
* COPD (FEV1 < 80%)
* Severe cardiovascular disease (NYHA > 3)
* Pregnancy
* Tobacco use
* Know or suspected difficulty with intubation
* Severe GERD or risk of aspiration

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antony Carrier-Boucher, MD, Principal Investigator — Laval University; Bussières S Jean, MD, Principal Investigator — Laval University
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

REFERENCES:
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Background] Juvin P, Lavaut E, Dupont H, Lefevre P, Demetriou M, Dumoulin JL, Desmonts JM. Difficult tracheal intubation is more common in obese than in lean patients. Anesth Analg. 2003 Aug;97(2):595-600. doi: 10.1213/01.ANE.0000072547.75928.B0. PMID 12873960
- [Background] Langeron O, Masso E, Huraux C, Guggiari M, Bianchi A, Coriat P, Riou B. Prediction of difficult mask ventilation. Anesthesiology. 2000 May;92(5):1229-36. doi: 10.1097/00000542-200005000-00009. PMID 10781266
- [Background] Tanoubi I, Drolet P, Donati F. Optimizing preoxygenation in adults. Can J Anaesth. 2009 Jun;56(6):449-66. doi: 10.1007/s12630-009-9084-z. Epub 2009 Apr 28. PMID 19399574
- [Background] Gambee AM, Hertzka RE, Fisher DM. Preoxygenation techniques: comparison of three minutes and four breaths. Anesth Analg. 1987 May;66(5):468-70. No abstract available. PMID 3578856
- [Background] Jense HG, Dubin SA, Silverstein PI, O'Leary-Escolas U. Effect of obesity on safe duration of apnea in anesthetized humans. Anesth Analg. 1991 Jan;72(1):89-93. doi: 10.1213/00000539-199101000-00016. PMID 1984382
- [Background] Damia G, Mascheroni D, Croci M, Tarenzi L. Perioperative changes in functional residual capacity in morbidly obese patients. Br J Anaesth. 1988 Apr;60(5):574-8. doi: 10.1093/bja/60.5.574. PMID 3377932
- [Background] Pelosi P, Croci M, Ravagnan I, Tredici S, Pedoto A, Lissoni A, Gattinoni L. The effects of body mass on lung volumes, respiratory mechanics, and gas exchange during general anesthesia. Anesth Analg. 1998 Sep;87(3):654-60. doi: 10.1097/00000539-199809000-00031. PMID 9728848
- [Background] Altermatt FR, Munoz HR, Delfino AE, Cortinez LI. Pre-oxygenation in the obese patient: effects of position on tolerance to apnoea. Br J Anaesth. 2005 Nov;95(5):706-9. doi: 10.1093/bja/aei231. Epub 2005 Sep 2. PMID 16143575
- [Background] Boyce JR, Ness T, Castroman P, Gleysteen JJ. A preliminary study of the optimal anesthesia positioning for the morbidly obese patient. Obes Surg. 2003 Feb;13(1):4-9. doi: 10.1381/096089203321136511. PMID 12630606
- [Background] Lane S, Saunders D, Schofield A, Padmanabhan R, Hildreth A, Laws D. A prospective, randomised controlled trial comparing the efficacy of pre-oxygenation in the 20 degrees head-up vs supine position. Anaesthesia. 2005 Nov;60(11):1064-7. doi: 10.1111/j.1365-2044.2005.04374.x. PMID 16229689
- [Background] Collins JS, Lemmens HJ, Brodsky JB, Brock-Utne JG, Levitan RM. Laryngoscopy and morbid obesity: a comparison of the "sniff" and "ramped" positions. Obes Surg. 2004 Oct;14(9):1171-5. doi: 10.1381/0960892042386869. PMID 15527629
- [Background] Levitan RM, Mechem CC, Ochroch EA, Shofer FS, Hollander JE. Head-elevated laryngoscopy position: improving laryngeal exposure during laryngoscopy by increasing head elevation. Ann Emerg Med. 2003 Mar;41(3):322-30. doi: 10.1067/mem.2003.87. PMID 12605198
- [Background] Coussa M, Proietti S, Schnyder P, Frascarolo P, Suter M, Spahn DR, Magnusson L. Prevention of atelectasis formation during the induction of general anesthesia in morbidly obese patients. Anesth Analg. 2004 May;98(5):1491-5, table of contents. doi: 10.1213/01.ane.0000111743.61132.99. PMID 15105237
- [Background] Cressey DM, Berthoud MC, Reilly CS. Effectiveness of continuous positive airway pressure to enhance pre-oxygenation in morbidly obese women. Anaesthesia. 2001 Jul;56(7):680-4. doi: 10.1046/j.1365-2044.2001.01374-3.x. PMID 11437771
- [Background] Gander S, Frascarolo P, Suter M, Spahn DR, Magnusson L. Positive end-expiratory pressure during induction of general anesthesia increases duration of nonhypoxic apnea in morbidly obese patients. Anesth Analg. 2005 Feb;100(2):580-584. doi: 10.1213/01.ANE.0000143339.40385.1B. PMID 15673897
- [Background] Delay JM, Sebbane M, Jung B, Nocca D, Verzilli D, Pouzeratte Y, Kamel ME, Fabre JM, Eledjam JJ, Jaber S. The effectiveness of noninvasive positive pressure ventilation to enhance preoxygenation in morbidly obese patients: a randomized controlled study. Anesth Analg. 2008 Nov;107(5):1707-13. doi: 10.1213/ane.0b013e318183909b. PMID 18931236
- [Background] Baraka AS, Hanna MT, Jabbour SI, Nawfal MF, Sibai AA, Yazbeck VG, Khoury NI, Karam KS. Preoxygenation of pregnant and nonpregnant women in the head-up versus supine position. Anesth Analg. 1992 Nov;75(5):757-9. doi: 10.1213/00000539-199211000-00018. PMID 1416130
- [Background] Lellouche F, Dionne S, Simard S, Bussieres J, Dagenais F. High tidal volumes in mechanically ventilated patients increase organ dysfunction after cardiac surgery. Anesthesiology. 2012 May;116(5):1072-82. doi: 10.1097/ALN.0b013e3182522df5. PMID 22450472
- [Result] Dixon BJ, Dixon JB, Carden JR, Burn AJ, Schachter LM, Playfair JM, Laurie CP, O'Brien PE. Preoxygenation is more effective in the 25 degrees head-up position than in the supine position in severely obese patients: a randomized controlled study. Anesthesiology. 2005 Jun;102(6):1110-5; discussion 5A. doi: 10.1097/00000542-200506000-00009. PMID 15915022
- [Derived] Couture EJ, Carrier-Boucher A, Provencher S, Tanoubi I, Marceau S, Bussieres JS. Effect of reverse Trendelenburg position and positive pressure ventilation on safe non-hypoxic apnea period in obese, a randomized-control trial. BMC Anesthesiol. 2023 Jun 8;23(1):198. doi: 10.1186/s12871-023-02128-7. PMID 37291541

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between September and December 2015 on the bariatric surgery ward during the preoperative assessment.
Pre-assignment Details: Files were evaluated in order to see if the patients met the inclusion criteria, if they had any exclusion criteria. Then the trial was explained to them and they could choose wether they wanted to participate or not.
  75 patients files were evaluated, 53 were solicitated, 3 refused to participate.
Groups:
- Reverse Trendelenburg and NIPPV: Table Position: Reverse Trendelenburg, Inclination of the whole table at 25 degrees from an horizontal plane, head up.
  NIPPV: 3 minutes of pre-oxygenation with 8 cm H2O positive pressure and 10 cm H2O PEEP. Trigger set at 1,5 L/min, mouth piece is used as a ventilatory interface
  Reverse Trendelenburg and NIPPV: Table Position: Reverse Trendelenburg, Inclination of the whole table at 25 degrees from an horizontal plane, head up.
  NIPPV: 3 minutes of pre-oxygenation with 8 cm H2O positive pressure and 10 cm H2O PEEP. Trigger set at 1,5 L/min, mouth piece is used as a ventilatory interface
Period: Overall Study
Arm/Group | Beach Chair (BC) and ZEEP | Reverse Trendelenburg and NIPPV
Started | 25 | 25
Completed | 24 | 24
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Saturometer malfunction | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beach Chair (BC) and ZEEP | Reverse Trendelenburg and NIPPV | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.1) | 40.8 (8.5) | 43.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 6 | 8 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 24 | 24 | 48
Weight (kg) [Mean (Standard Deviation); unit: kilogram] | 129 (20.8) | 131.7 (11.1) | 130.4 (10.2)
Height (m) [Mean (Standard Deviation); unit: centimeters] | 1.6 (0.1) | 1.7 (0.1) | 1.7 (0.1)
BMI (m/kg2) [Mean (Standard Deviation); unit: kilogram per meter square] | 47.3 (5.2) | 47.9 (6.3) | 47.6 (5.7)
Waist circumference (cm) [Mean (Standard Deviation); unit: centimeters] | 113.5 (14.7) | 138.4 (15) | 136.1 (14.7)
Hip circumference (cm) [Mean (Standard Deviation); unit: centimeters] | 136.4 (11.1) | 142.8 (14.8) | 139.6 (13.3)
Waist:hip ratio [Mean (Standard Deviation); unit: ratio] | 1.0 (0.1) | 1.0 (0.1) | 1.0 (0.1)
Neck Circumference [Mean (Standard Deviation); unit: centimeters] | 44.9 (4.8) | 43.9 (5.9) | 44.4 (5.3)
FEV1 (liters) [Mean (Standard Deviation); unit: liters] — Population: We evaluated the FEV1 of the patients we had in the files
  liters
    number analyzed (Participants) | 15 | 19 | 34
    (all) | 2.8 (0.6) | 2.9 (0.8) | 2.9 (0.7)
Sleep apnea Dx (n) [Number; unit: participants] | 11 | 12 | 23
CPAP [Number; unit: participants] | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Non Hypoxic Apnea Time
Description: Change of Non-hypoxic apnea time in obese patient during a General Anesthesia induction, as a result of different pre-oxygenation position and ventilation mode; 1-Beach Chair and No positive pressure ventilation, 2-Reverse Trendelenburg and positive pressure ventilation and PEEP. End of measure time frame is 5 minutes after intubation
Time Frame: After a 3 minutes pre-oxygenation period
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Beach Chair (BC) and ZEEP | Reverse Trendelenburg and NIPPV
Number analyzed (Participants) | 24 | 24
seconds | 216.7 (42.3) | 258.2 (55.1)
Statistical Analysis 1: Comparison: Beach Chair (BC) and ZEEP vs Reverse Trendelenburg and NIPPV; We calculated our sample size using data from EPO2: PV study (Couture: simultaneous submitted manuscript), where we found a difference in the FRC of 21% between reverse Trendelenburg with non-invasive positive pressure ventilation and beach chair position without positive pressure ventilation. Assuming there would be a difference of 21% in the apnea time, with a type I error of 5% and power of 80%, a total of 17 patients by group was needed; Test type: Superiority or Other; p = 0.005, ANOVA

2. Secondary Outcome: Time to Expired Oxygen Fraction > 0,9
Description: Evaluation of time needed to obtain an expired fraction of oxygen of > 0,9 in the two groups during the pre-oxygenation
Time Frame: During the pre-oxygenation period
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Beach Chair (BC) and ZEEP | Reverse Trendelenburg and NIPPV
Number analyzed (Participants) | 24 | 24
seconds | 145.3 (40.8) | 85.1 (47.8)
Statistical Analysis 1: Comparison: Beach Chair (BC) and ZEEP vs Reverse Trendelenburg and NIPPV; Test type: Superiority or Other; p < 0.0001, ANOVA

3. Secondary Outcome: Maximum Expired Fraction of Oxygen Obtained
Description: Evaluation of the maximum expired oxygen fraction obtained in the two groups
Time Frame: After 3 minutes of pre-oxygenation
Measure: Mean (Standard Deviation); unit: Maximum expired fraction of oxygen obtai
Arm/Group | Beach Chair (BC) and ZEEP | Reverse Trendelenburg and NIPPV
Number analyzed (Participants) | 24 | 24
Maximum expired fraction of oxygen obtai | 0.89 (0.01) | 0.91 (0.01)
Statistical Analysis 1: Comparison: Beach Chair (BC) and ZEEP vs Reverse Trendelenburg and NIPPV; Test type: Superiority or Other; p = 0.0003, ANOVA

4. Secondary Outcome: Minimum Arterial Saturation of Oxygen Obtained
Description: Evaluation of the minimal saturation obtained after the resumption of the ventilation
Time Frame: After the end of the Non-hypoxic apnea time
Population: One patient missing in the BC group
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Beach Chair (BC) and ZEEP | Reverse Trendelenburg and NIPPV
Number analyzed (Participants) | 23 | 24
percent | 83.6 (0.9) | 85.3 (4.5)
Statistical Analysis 1: Comparison: Beach Chair (BC) and ZEEP vs Reverse Trendelenburg and NIPPV; Test type: Superiority or Other; p = 0.9, ANOVA

5. Secondary Outcome: Time to 97% Saturation
Time Frame: Evaluation of the time needed to the beginning of the ventilation to the moment where the saturation is 97%
Population: 4 values missing in the BC group and 5 values missing in RT group.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Beach Chair (BC) and ZEEP | Reverse Trendelenburg and NIPPV
Number analyzed (Participants) | 21 | 20
seconds | 88.4 (17.3) | 68 (10.6)
Statistical Analysis 1: Comparison: Beach Chair (BC) and ZEEP vs Reverse Trendelenburg and NIPPV; Test type: Superiority or Other; p = 0.03, ANOVA

6. Secondary Outcome: Hemodynamic Changes
Description: Evaluation of the changes in vital signs during and after the pre-oxygenation phase in the two combinations of position and ventilation mode
Time Frame: From the beginning of the pre-oxygenation to the end of the protocol
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 15 minutes
Description: the patients were not followed after the research protocol, after the patient oxygen saturation reached 97 %, the protocol ended and did not follow the patients afterwards
Arm/Group | Beach Chair (BC) and ZEEP | Reverse Trendelenburg and NIPPV
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
The main limitation of this study is that we did not compare the position and ventilation mode separately. The reason why we decided to do it as a bundle of interventions was that we wanted to minimize the number of patients exposed to the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No